CLINICAL TRIAL: NCT00484276
Title: NGR010: A Phase II Study of NGR-hTNF Administered as Single Agent Every 3 Weeks or Weekly in Patients Affected by Advanced or Metastatic Malignant Pleural Mesothelioma Previously Treated With no More Than One Systemic Therapeutic Regimen
Brief Title: Study of NGR-hTNF as Single Agent in Patients Affected by Advanced or Metastatic Malignant Pleural Mesothelioma
Acronym: NGR010
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGR010; 2006-005993-39 (EudraCT Number)
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: NGR-hTNF; malignant pleural mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — tumor necrosis factor-alpha, CNGRC fusion protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NGR-hTNF (Experimental): NGR-hTNF: 0.8 mcg/m² as 60 minutes intravenous infusion every 3 weeks or weekly
  Interventions: Drug: NGR-hTNF

INTERVENTIONS:
Drug: NGR-hTNF — iv q3W or q1W 0.8 mcg/sqm NGR-hTNF

SUMMARY:
The main objective of the trial is to document the progression free survival (PFS) in advanced or metastatic malignant pleural mesothelioma patients treated with NGR-hTNF as single agent.

Safety will be established by clinical and laboratory assessment according to NCI-CTC criteria.

DETAILED DESCRIPTION:
This is a phase II, open-label, non-randomized study that will be conducted in patients affected by advanced or metastatic malignant pleural mesothelioma previously treated with no more than one systemic therapeutic regimen , that will be conducted using Simon's two-stage design method.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years affected by malignant pleural mesothelioma previously treated with no more than one systemic therapeutic regimen
* Histologically or cytological confirmed malignant pleural mesothelioma of any of the following subtype: epithelial, sarcomatous, mixed
* Prior intrapleural cytotoxic agents including bleomycin not considered systemic chemotherapy
* ECOG Performance status 0 - 2
* Adequate baseline bone marrow, hepatic and renal function, defined as follows:

  * Neutrophils > 1.5 x 10^9/L and platelets > 100 x 10^9/L
  * Bilirubin < 1.5 x ULN
  * AST and/or ALT < 2.5 x ULN in absence of liver metastasis
  * AST and/or ALT < 5 x ULN in presence of liver metastasis
  * Serum creatinine < 1.5 x ULN
* Absence of any conditions in which hypervolemia and its consequences (e.g. increased stroke volume, elevated blood pressure) or haemodilution could represent a risk for the patient (take as reference "Technical data sheet human albumin" specifically used in Pharmacy Department for NGR-hTNF dilution)
* Patients may have had prior therapy providing the following conditions are met:

  * Chemotherapy and radiotherapy: wash-out period of 28 days
  * Surgery: wash-out period of 14 days
* Normal cardiac function and absence of uncontrolled hypertension
* Patients must give written informed consent to participate in the study

Exclusion Criteria:

* Concurrent anticancer therapy
* Patients may not receive any other investigational agents while on study
* Clinical signs of CNS involvement
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Known hypersensitivity/allergic reaction to human albumin preparations or to any of the excipients
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation. Patients - both males and females - with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Antitumor activity defined as progression free survival (PFS) | during the study
  Defined as the time from the date of randomization until disease progression, or death

SECONDARY OUTCOMES:
Tumor Growth Control Rate (TGCR) | Every 6 weeks during study treatment and every 6 weeks during the follow-up before PD
  Evaluated according to modified RECIST criteria for Malignant Pleural Mesothelioma
Overall survival (OS) | from the randomization until to the date of patient death or discontinuation from the study
  Defined as the time from the date of randomization until the date of death due to any cause or the last date the patient was known to be alive
Experimental Imaging Study (DCE-MRI) | During the treatment
  To document possible modifications on vessels permeability by imaging techniques
Cmax of NGR-hTNF in patients treated with weekly schedule | During the treatment
  to evaluate Cmax of NGR-hTNF administered weekly
AUC(tau) of NGR-hTNF in patients treated with weekly schedule | During the treatment
  to evaluate AUC(tau) of NGR-hTNF administered weekly
Safety according to NCI-CTCAE criteria (version 3) | During the treatment and during the follow-up
  To evaluate safety profile related to NGR-hTNF

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (4):
- Italy (4):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Fondazione San Raffaele del Monte Tabor, Milan
  - Istituto Europeo Oncologico, Milan
  - Istituto Nazionale dei Tumori, Milan

REFERENCES:
- [Result] Gregorc V, Zucali PA, Santoro A, Ceresoli GL, Citterio G, De Pas TM, Zilembo N, De Vincenzo F, Simonelli M, Rossoni G, Spreafico A, Grazia Vigano M, Fontana F, De Braud FG, Bajetta E, Caligaris-Cappio F, Bruzzi P, Lambiase A, Bordignon C. Phase II study of asparagine-glycine-arginine-human tumor necrosis factor alpha, a selective vascular targeting agent, in previously treated patients with malignant pleural mesothelioma. J Clin Oncol. 2010 May 20;28(15):2604-11. doi: 10.1200/JCO.2009.27.3649. Epub 2010 Apr 20. PMID 20406925